CLINICAL TRIAL: NCT06803238
Title: Procedural Mitral Isthmus Block Durability After Pulsed-Field Ablation in Patients with Non-Paroxysmal Atrial Fibrillation
Acronym: FARA Block
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: FARA Block
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; catheter ablation; pulsed-field ablation; mitral isthmus
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Mitral isthmus is one of the targets for the catheter ablation of non-paroxysmal atrial fibrillation (AF), in which pulmonary veins isolation alone is not deemed sufficient. Typically, lateral mitral isthmus ablation line is performed from the mitral annulus to the ostium of the left inferior pulmonary vein or to the posterior base of the left atrial appendage. When conduction block across the mitral isthmus is achieved, the standard practice using radiofrequency energy is to wait 20 minutes to verify durability of the conduction block.

Currently, there is an increase in procedures performed using pulsed-field energy (PF). The procedure is in most centers terminated immediately after the energy is delivered, and, unlike radiofrequency energy procedures, there is no waiting period to see if the conduction through the ablation lines returns. However return of conduction across the mitral isthmus has been described during reablation procedures performed for clinical recurrence of arrhythmia (perimitral flutter or atrial fibrillation).

The presented study is a follow-up of previous work, which included 30 patients with non-paroxysmal AF, who underwent PF ablation including mitral isthmus ablation as part of the procedure. Ablation of the mitral isthmus was performed by repeated series of 9 PF energy applications. After each series a waiting period of 20 minutes followed. In case of recurrence of conduction, another series of 9 PF applications was delivered followed by a new waiting period. In the cases of reconduction after the 3rd series, one last series of PF applications was performed, where the number of applications was left at the discretion of the operator, where the total number of applications delivered to the mitral isthmus could not exceed 50. We found that although conduction block on the mitral isthmus was achieved in 90 % of patients after all series, it was only in 33,3 % of patients after the first series. Repeated waiting and multiple ablation series prolonged the procedure unnecessarily. On the other hand, a very high number of pulsed-field energy applications applied initially could be associated with a risk of hemolysis. So far, the number of PF applications up to 80-100 were demonstrated to be safe.

This present study aims to determine whether increasing the number of applications in the first series delivered to the mitral isthmus will be associated with faster and durable achievement of conduction block across the mitral isthmus.

A total of 40 patients with symptomatic non-paroxysmal AF, indicated for catheter ablation according to current guidelines, will be included. Patients with previous left atrial ablation, presenting left ventricular dysfunction with LV EF < 30%, as well as patients at high risk of prolonged analgosedation (i.g. history of severe COPD, treated OSA) will be excluded. The procedure will be performed according to the standards of our center, i.e. pulmonary veins isolation, left atrial posterior wall ablation and mitral isthmus ablation will be performed. All procedures will be performed under analgosedation or general anesthesia controlled by an anesthesiologist. All ablations will be made using PF energy (system FARAPULSE, Boston sci., USA) and under control of intracardiac echocardiography. In contrast to previous work, a total of 20 applications of PF energy will be administered to the mitral isthmus in the first series of ablation. A waiting period of 20 minutes will follow, during which the conduction block across the mitral isthmus will be verified by assessment of the activation sequence on the decapolar catheter in the coronary sinus when pacing from the base of the left atrial appendage and by assessment of the activation of the left atrial appendage when pacing from the distal coronary sinus (or by differential pacing in case of uncertainity). If there is no recurrence of conduction across the mitral isthmus within 20 min, the procedure will be terminated. If recurrence does occur, a second series of 20 PF energy applications will be administered and another 20-minute waiting period will be initiated. In the case of reconduction after the 2nd series, one last optional ablation series will be delivered at the discretion of the operator. For safety reasons, the total waiting time will be 40 minutes and the total number of PF energy applications to the mitral isthmus will be limited to 50 (in the third series, only 10 applications can be delivered). After the procedure, the catheters and sheaths will be withdrawn and the site of puncture fixed with Z suture. All patients will receive 1000 mL of saline postproceduraly and will be endouredged to drink sufficient amount of fluids on the day after the procedure. Renal function (BUN, creatinine) will be assessed on the following day after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with symptomatic non-paroxysmal atrial fibrillation indicated for catheter ablation according to the current guidelines

Exclusion Criteria:

* Contraindication to catheter ablation according to the current guidelines
* previous left atrial ablation
* left ventricular dysfunction with LV EF < 30%
* Patients at high risk of prolonged analgosedation, e.g. history of severe COPD (stage 3 or 4), obstructive sleep apnea on treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for catheter ablation of non paroxysmal AF by referring cardiologists and from arrythmology clinic
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Mitral isthmus block durability after 1 series of PF applications | 20 minutes after last PF application
  Acute mitral isthmus conduction block sustained for a waiting period of 20 minutes after 1 series of 20 PF applications

SECONDARY OUTCOMES:
Overall mitral isthmus block durability | 20 minutes after last PF application of last ablation series
  Overall acute mitral isthmus conduction block achieved by the protocol-defined ablation (of up to 3 ablation series of up to 50 PF applications) and sustained for a waiting period of 20 minutes

REFERENCES:
- [Derived] Hornof J, Hozman M, Herman D, Romanenko O, Hassouna S, Vesela J, Filipcova V, Poviser L, Karch J, Hozmanova J, Znojilova L, Molova A, Penkava V, Osmancik P. Acute Efficacy of Pulsed-Field Ablation of the Mitral Isthmus Using a Pentaspline Catheter and Two Different Ablation Settings. J Cardiovasc Electrophysiol. 2025 Dec 27. doi: 10.1111/jce.70236. Online ahead of print. PMID 41456097